CLINICAL TRIAL: NCT00620282
Title: The Effect of Liraglutide on Endothelial Function in Subjects With Type 2 Diabetes Mellitus: A 12-week Randomized, Double-blind, Placebo-controlled, Parallel-group, Single-center Trial With an Open-label Glimepiride Arm
Brief Title: The Effect of Liraglutide on Endothelial Function in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN2211-1799
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Results first posted 2011-06-15 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Liraglutide; glimepiride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lira 1.8 (Experimental): Liraglutide 1.8 mg administered subcutaneously, once-daily, weeks 0-12 (100 uL/day, week 1; 200 uL/day, week 2; 300 uL/day, week 3-12)
  Interventions: Drug: liraglutide
- Placebo (Placebo Comparator): Placebo administered subcutaneously, once-daily, weeks 0-12 (100 uL/day, week 1; 200 uL/day, week 2; 300 uL/day, week 3-12)
  Interventions: Drug: placebo
- Glimepiride (Active Comparator): Glimepiride 4 mg administered orally, once-daily, open-label, weeks 0-12
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: liraglutide — Stepwise dose increase, s.c. (under the skin) injection, once daily
  Arms: Lira 1.8
Drug: placebo — Liraglutide placebo, stepwise dose increase, s.c. (under the skin) injection, once daily
  Arms: Placebo
Drug: glimepiride — Tablets, 1 - 4 mg daily
  Arms: Glimepiride

SUMMARY:
This trial is conducted in the United States of America (USA). The purpose of the trial is to assess the effect of liraglutide on forearm blood flow in subjects with type 2 diabetes who are on diet and lifestyle changes or treated with metformin alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Diet and lifestyle changes or metformin monotherapy for at least three months
* HbA1c (glycosylated haemoglobin) 6.5-9.0% (both inclusive)
* Body Mass Index (BMI) less than or equal to 40 kg/m^2

Exclusion Criteria:

* Previous treatment with insulin (except for short term treatment with insulin in connection with intercurrent illness, at the discretion of the Investigator)
* Previous treatment with glucagon-like peptide-1 (GLP-1) analogues/mimetics, including treatment in a clinical trial
* Treatment with any oral hypoglycaemic agents other than metformin in a period of 3 months prior to screening
* Current smoker or history of smoking within 6 months prior to screening
* Evidence of overt cardiovascular disease (documented coronary heart disease, class II-IV congestive heart failure, cerebrovascular disease, or peripheral vascular disease)
* Abnormal, clinically significant exercise stress electrocardiogram (ECG) test, as judged by the Investigator
* Known retinopathy or maculopathy requiring acute treatment, as judged by the Investigator
* Known autonomic neuropathy, as judged by the Investigator
* Initiation or change (dose or treatment regimen) in concomitant blood pressure-lowering or lipid-lowering medication within 4 weeks prior to screening
* Systolic blood pressure more than or equal to 140 mmHg and/or diastolic blood pressure more than or equal to 90 mmHg

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Rochester, Minnesota, United States

REFERENCES:
- [Result] Alves C, Batel-Marques F, Macedo AF. A meta-analysis of serious adverse events reported with exenatide and liraglutide: acute pancreatitis and cancer. Diabetes Res Clin Pract. 2012 Nov;98(2):271-84. doi: 10.1016/j.diabres.2012.09.008. Epub 2012 Sep 23. PMID 23010561
- [Result] Nandy D, Johnson C, Basu R, Joyner M, Brett J, Svendsen CB, Basu A. The effect of liraglutide on endothelial function in patients with type 2 diabetes. Diab Vasc Dis Res. 2014 Nov;11(6):419-30. doi: 10.1177/1479164114547358. Epub 2014 Sep 11. PMID 25212693
- [Result] Jensen TM, Saha K, Steinberg WM. Is there a link between liraglutide and pancreatitis? A post hoc review of pooled and patient-level data from completed liraglutide type 2 diabetes clinical trials. Diabetes Care. 2015 Jun;38(6):1058-66. doi: 10.2337/dc13-1210. Epub 2014 Dec 12. PMID 25504028
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at one site in the United States of America (USA).
Period: Overall Study
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Started | 16 | 16 | 17
Completed | 16 | 14 | 16
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Arterial line unable to be placed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lira 1.8 | Placebo | Glimepiride | Total
Number analyzed (Participants) | 16 | 16 | 17 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (9.0) | 60.3 (7.3) | 57.7 (5.3) | 58.5 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 10 | 10 | 11 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 16 | 16 | 17 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 16 | 16 | 17 | 49
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 5.3 (4.1) | 8.4 (4.6) | 6.8 (8.1) | 6.8 (6.0)
Previous Anti-diabetic Treatment [Number; unit: participants]
  Diet/Exercise | 2 | 1 | 2 | 5
  Metformin | 14 | 15 | 15 | 44
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 32.7 (4.5) | 31.6 (4.2) | 31.1 (4.9) | 31.8 (4.5)
Body Weight [Mean (Standard Deviation); unit: kg] | 95.09 (13.12) | 90.63 (13.47) | 91.99 (13.97) | 92.56 (13.38)
Glycosylated Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of total haemoglobin] | 7.2 (0.5) | 7.0 (0.5) | 7.3 (0.5) | 7.2 (0.5)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 160.8 (31.2) | 145.2 (20.1) | 163.3 (33.3) | 156.6 (29.4)
Total Cholesterol (TC) [Mean (Standard Deviation); unit: mg/dL] | 170.2 (34.4) | 157.5 (32.0) | 160.2 (24.1) | 162.6 (30.2)
Low density lipoprotein (LDL-C) [Mean (Standard Deviation); unit: mg/dL] | 102.8 (31.3) | 92.5 (23.5) | 94.1 (18.4) | 96.4 (24.8)
High density lipoprotein (HDL-C) [Mean (Standard Deviation); unit: mg/dL] | 39.6 (10.0) | 39.2 (7.5) | 43.5 (10.3) | 40.8 (9.4)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] | 165.8 (72.9) | 145.9 (57.5) | 141.4 (67.4) | 150.8 (65.7)
Tumor necrosis factor-alpha (TNF-alpha) [Mean (Standard Deviation); unit: pg/mL] | 2.1 (1.5) | 1.4 (0.8) | 1.4 (0.5) | 1.6 (1.0)

OUTCOME MEASURES:

1. Primary Outcome: Change in Acetylcholine (ACh)-Mediated Forearm Blood Flow (FBF)
Description: Assessed endothelial function by measuring the change in ACh-mediated FBF at euglycemia (90 mg/dL) using forearm venous occlusion plethysmography (VOP) technique. Unit of Measure refers to volume of blood (mL) per 100 mL of forearm tissue per minute.
Time Frame: week 0, week 12
Population: The ANCOVA full analysis set (FAS) includes all randomised subjects for whom data points could be collected at end of trial.
Measure: Least Squares Mean (Standard Error); unit: mL/100 mL/min
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mL/100 mL/min | 4.244 (2.551) | -3.187 (2.758) | 2.164 (2.568)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in Ach-mediated FBF from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline FBF as a covariate; Test type: Superiority or Other; p = 0.0549, ANCOVA — 2-sided significance level of 5%; Least squares mean = 7.43, 95% CI [-0.164 to 15.025]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.5681, ANCOVA — 2-sided significance level of 5%; Least squares mean = 2.08, 95% CI [-5.215 to 9.375]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.1668, ANCOVA — 2-sided significance level of 5%; Least squares mean = 5.35, 95% CI [-2.323 to 13.024]

2. Secondary Outcome: Change in Sodium Nitroprusside (SNP)-Mediated Forearm Blood Flow (FBF)
Description: Assessed endothelial function by measuring the change in SNP-mediated FBF at euglycemia (90 mg/dL) using forearm venous occlusion plethysmography (VOP) technique. Unit of Measure refers to volume of blood (mL) per 100 mL of forearm tissue per minute.
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL/100 mL/min
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mL/100 mL/min | 3.455 (2.681) | -1.044 (2.893) | 2.746 (2.67)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in SNP-mediated FBF from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline FBF as a covariate; Test type: Superiority or Other; p = 0.2648, ANCOVA — 2-sided significance level of 5%; Least squares mean = 4.499, 95% CI [-3.535 to 12.534]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.8518, ANCOVA — 2-sided significance level of 5%; Least squares mean = 0.709, 95% CI [-6.904 to 8.322]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.3435, ANCOVA — 2-sided significance level of 5%; Least squares mean = 3.79, 95% CI [-4.194 to 11.774]

3. Secondary Outcome: Change in HbA1c (Glycosylated Haemoglobin A1c)
Description: Percentage point change in HbA1c
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of total haemoglobin
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
percentage of total haemoglobin | -0.629 (0.109) | -0.094 (0.121) | -0.552 (0.112)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in HbA1c from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HbA1c as a covariate; Test type: Superiority or Other; p = 0.0023, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.536, 95% CI [-0.868 to -0.203]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.6207, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.077, 95% CI [-0.391 to 0.236]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0098, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.458, 95% CI [-0.8 to -0.116]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG)
Description: Change in FPG
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mg/dL | -41.672 (3.643) | -6.067 (4.079) | -32.019 (3.708)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in FPG from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline FPG as a covariate; Test type: Superiority or Other; ANCOVA — 2-sided significance level of 5%; Least squares mean = -35.605, 95% CI [-46.797 to -24.413]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.0677, ANCOVA — 2-sided significance level of 5%; Least squares mean = -9.653, 95% CI [-20.041 to 0.736]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; ANCOVA — 2-sided significance level of 5%; Least squares mean = -25.952, 95% CI [-37.429 to -14.475]

5. Secondary Outcome: Change in Mean Postprandial Glucose (PPG) Based on Self-measured 7-point Plasma Glucose Profiles
Description: The 7-point profile included plasma glucose measurements at the following time points: before each main meal (breakfast, lunch and dinner), 90 minutes after the start of each main meal (breakfast, lunch and dinner) and at bedtime.
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 13 | 10 | 14
mg/dL | -32.175 (9.104) | -20.304 (10.619) | -35.99 (8.673)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in PPG from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline PPG as a covariate; Test type: Superiority or Other; p = 0.4121, ANCOVA — 2-sided significance level of 5%; Least squares mean = -11.871, 95% CI [-40.943 to 17.201]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7622, ANCOVA — 2-sided significance level of 5%; Least squares mean = 3.815, 95% CI [-21.618 to 29.247]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.2651, ANCOVA — 2-sided significance level of 5%; Least squares mean = -15.686, 95% CI [-43.838 to 12.466]

6. Secondary Outcome: Change in Body Weight
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 17
kg | -1.821 (0.455) | -0.293 (0.486) | 1.038 (0.441)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in body weight from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline body weight as a covariate; Test type: Superiority or Other; p = 0.0268, ANCOVA — 2-sided significance level of 5%; Least squares mean = -1.528, 95% CI [-2.873 to -0.184]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; ANCOVA — 2-sided significance level of 5%; Least squares mean = -2.859, 95% CI [-4.139 to -1.579]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0486, ANCOVA — 2-sided significance level of 5%; Least squares mean = 1.331, 95% CI [0.0090 to 2.653]

7. Secondary Outcome: Fasting Lipid Profile - Change in Total Cholesterol (TC)
Description: Change in TC
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mg/dL | 2.006 (5.274) | 4.243 (5.597) | 0.094 (5.239)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in TC from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline TC as a covariate; Test type: Superiority or Other; p = 0.7736, ANCOVA — 2-sided significance level of 5%; Least squares mean = -2.237, 95% CI [-17.829 to 13.354]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.7993, ANCOVA — 2-sided significance level of 5%; Least squares mean = 1.912, 95% CI [-13.168 to 16.991]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.5903, ANCOVA — 2-sided significance level of 5%; Least squares mean = -4.149, 95% CI [-19.582 to 11.284]

8. Secondary Outcome: Fasting Lipid Profile - Change in LDL-C
Description: Change in LDL-C
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mg/dL | 1.243 (4.294) | -2.459 (4.551) | -1.529 (4.275)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in LDL-C from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline LDL-C as a covariate; Test type: Superiority or Other; p = 0.5583, ANCOVA — 2-sided significance level of 5%; Least squares mean = 3.702, 95% CI [-8.96 to 16.365]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.6517, ANCOVA — 2-sided significance level of 5%; Least squares mean = 2.773, 95% CI [-9.537 to 15.082]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.8822, ANCOVA — 2-sided significance level of 5%; Least squares mean = 0.929, 95% CI [-11.646 to 13.505]

9. Secondary Outcome: Fasting Lipid Profile - Change in HDL-C
Description: Change in HDL-C
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mg/dL | 0.393 (1.053) | 0.562 (1.133) | 1.116 (1.074)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in HDL-C from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline HDL-C as a covariate; Test type: Superiority or Other; p = 0.9131, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.169, 95% CI [-3.273 to 2.935]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.6362, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.723, 95% CI [-3.785 to 2.339]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.7283, ANCOVA — 2-sided significance level of 5%; Least squares mean = 0.554, 95% CI [-2.643 to 3.751]

10. Secondary Outcome: Fasting Lipid Profile - Change in Triglycerides (TG)
Description: Change in TG
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 14 | 16
mg/dL | -8.163 (13.471) | 28.546 (14.282) | -4.377 (13.399)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in TG from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline TG as a covariate; Test type: Superiority or Other; p = 0.0694, ANCOVA — 2-sided significance level of 5%; Least squares mean = -36.709, 95% CI [-76.467 to 3.048]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.844, ANCOVA — 2-sided significance level of 5%; Least squares mean = -3.786, 95% CI [-42.373 to 34.801]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 10, analysis 1]; Test type: Superiority or Other; p = 0.0994, ANCOVA — 2-sided significance level of 5%; Least squares mean = -32.923, 95% CI [-72.353 to 6.507]

11. Secondary Outcome: Biomarkers of Cardiovascular Risk - Change in TNF-alpha
Description: Change in TNF-alpha
Time Frame: week 0, week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/mL
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 12 | 10 | 12
pg/mL | -0.024 (0.232) | 0.397 (0.25) | -0.0050 (0.231)
Statistical Analysis 1: Comparison: Lira 1.8 vs Placebo; Change in TNF-alpha from baseline to end of treatment at 12 weeks was analysed using an analysis of covariance (ANCOVA) model with treatment as a fixed effect and baseline TNF-alpha as a covariate; Test type: Superiority or Other; p = 0.2282, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.42, 95% CI [-1.118 to 0.278]
Statistical Analysis 2: Comparison: Lira 1.8 vs Glimepiride; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.9569, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.018, 95% CI [-0.697 to 0.661]
Statistical Analysis 3: Comparison: Placebo vs Glimepiride; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.2465, ANCOVA — 2-sided significance level of 5%; Least squares mean = -0.402, 95% CI [-1.097 to 0.293]

12. Secondary Outcome: Haematology and Biochemistry Tests - Number of Subjects With Blood Urea Nitrogen (BUN) Values Outside Reference Range
Description: Number of subjects with serum BUN values outside reference range at Week 0 and Week 12, respectively. Reference range: Female (lower value 6.000 mg/dL, upper value 21.000 mg/dL) Male (lower value 8.000 mg/dL, upper value 25.000 mg/dL).
Time Frame: week 0, week 12
Population: Safety population included all subjects exposed to at least one dose of the drug or who underwent at least one venous occlusion plethysmography (VOP) procedure.
Measure: Number; unit: participants
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 16 | 17
participants
  Week 0 | 1 | 0 | 1
  Week 12 | 1 | 2 | 0

13. Secondary Outcome: Haematology and Biochemistry Tests - Number of Subjects With Creatinine Values Outside Reference Range
Description: Number of subjects with serum creatinine values outside reference range at Week 0 and Week 12, respectively. Reference range: Female (lower value 0.600 mg/dL, upper value 1.100 mg/dL) Male (lower value 0.800 mg/dL, upper value 1.300 mg/dL).
Time Frame: week 0, week 12
Population: as for outcome 12
Measure: Number; unit: participants
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 16 | 17
participants
  Week 0 | 1 | 3 | 5
  Week 12 | 1 | 2 | 2

14. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Total number of hypoglycaemic episodes occurring from week 0 to week 12. Hypoglycaemic episodes were defined as major, minor, or symptoms only. Major if the subject was unable to treat her/himself and either plasma glucose was below 56 mg/dL or symptoms were reversed after food intake or glucagon/intravenous glucose administration. Minor if subject was able to treat her/himself and plasma glucose was below 56 mg/dL. Symptoms only if subject was able to treat her/himself and with no plasma glucose measurement or plasma glucose higher than or equal to 56 mg/dL.
Time Frame: weeks 0-12
Population: as for outcome 12
Measure: Number; unit: episodes
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Number analyzed (Participants) | 16 | 16 | 17
episodes
  Major | 0 | 0 | 0
  Minor | 1 | 0 | 10
  Symptoms Only | 3 | 0 | 4

ADVERSE EVENTS:
Time Frame: The adverse events were collected from week 0 to week 12.
Description: The full safety analysis set is all subjects exposed to at least one dose of the drug or who underwent at least one venous occlusion plethysmography (VOP) procedure.
Arm/Group | Lira 1.8 | Placebo | Glimepiride
Serious Adverse Events (participants affected / at risk) | 0/16 | 1/16 | 0/17
Other Adverse Events (participants affected / at risk) | 11/16 | 9/16 | 5/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 (N=16) | Placebo (N=16) | Glimepiride (N=17)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lira 1.8 (N=16) | Placebo (N=16) | Glimepiride (N=17)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Parotid Duct Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Catheter Site Haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle Disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk reserves the right to not release data until specified milestones (e.g. when clinical trial report is available), including right to not release interim results because such action can invalidate results of the entire trial. At trial end, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.